CLINICAL TRIAL: NCT03178500
Title: Clomiphene Citrate Stair-step Protocol for Ovulation Induction in Women With Polycystic Ovarian Syndrome: A Randomized Clinical Trial
Brief Title: Clomiphene Citrate Stair-Step Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, ADEL SHAFIK SALAH EL-DIN, Assistant professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAIRSTEP TRIAL
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Polycystic Ovary
Keywords: clomiphene citrate; stair- step; poly cystic ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional (Experimental): Clomiphene citrate (50mg) will be given for 5 days (days 3-7). Transvaginal ultrasound from 9th-20th every other day if ovulation occur the patient will be excluded. If no ovulation, we will wait for the next menses and increase the dose to (100mg). if no ovulation occurred increase the dose to (150mg) in the next cycle if no ovulation increase the dose to (200mg) TVUS from 9th-20th ovary other day. If no ovulation we will wait for next cycle and increase the dose to (250mg) and so till 6 cycles.
  Interventions: Drug: Clomiphene Citrate 50mg
- Stair step protocol (Experimental): If there is no response (no follicle >10mm), so, (100mg) clomiphene will be initiated immediately for 5 days and ultrasound will be repeated 1 week after the first ultrasound. If there is no response, (150mg) clomiphene will be initiated immediately for another 5 days and TV/US will be performed 1 week after the second TV/US
  Interventions: Drug: Clomiphene Citrate 50mg

INTERVENTIONS:
Drug: Clomiphene Citrate 50mg — stair-step clomiphene adminstration

SUMMARY:
A RCT will be conducted to compare the traditional clomiphene citrate regimens for ovulation induction with the stair-step protocol. Sixty women will be included after obtaining their written informed consent and will be randomized into either of the 2 groups.

DETAILED DESCRIPTION:
This study is a randomized clinical trial (RCT) will be conducted in Ain Shams University maternity hospital at infertility clinic within a period of 6-8 months.

All patient are previously diagnosed as PCOs according to the Rotterdam conference of 2003.

All patients will be devided according to computer based program into two groups First group: Patients with traditional protocol

Traditional protocol:

Clomiphene citrate (clomid) (50mg) will be given for 5 days (days 3-7). Transvaginal ultrasound from 9th-20th every other day if ovulation occur the patient will be excluded if no ovulation, we will wait for the next menses and increase the dose to (100mg). if no ovulation occurred increase the dose to (150mg) in the next cycle if no ovulation increase the dose to (200mg) TVUS from 9th-20th ovary other day. If no ovulation we will wait for next cycle and increase the dose to (250mg) and so till 6 cycles .

Second group: Patient with stair step protocol Follicular development will be monitored using transvaginal ultrasound at 11-14 day after (50mg) clomiphene for 5 days if there is no response (no follicle >10mm), so, (100mg) clomiphene will be initiated immediately for 5 days and ultrasound will be repeated 1 week after the first ultrasound. If there is no response, (150mg) clomiphene will be initiated immediately for another 5 days and TV/US will be performed 1 week after the second TV/US .

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-35 years.

  * Body mass index (BMI/m2) 26-35 kg/m2
  * Normal hystrosalpingogram (HSG).
  * Normal Prolactin level.
  * Normal semen analysis.

Exclusion Criteria:

* - They underwent ovarian drilling.
* Other factors infertility.
* AUTOimmune diseases as thyroid disorders and systemic lupus erythematosus.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the ovulation by transvaginal ultrasound | 20 days
  * Follicle suddenly disappears or regresses in size.
  * Irregular margins.
  * Intra follicular echos. Follicle suddenly becomes more echogenic.
  * Free fluid in pouch of douglas.

SECONDARY OUTCOMES:
time to achieve ovulation | 20 days
  time for ovulation to occur
dose of clomiphene to achieve ovulation | 20 days
  the total dose of clomiphene used till ovulation

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Salah El-Din, MD, Study Director — Assistant Proffesor
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided